CLINICAL TRIAL: NCT03759327
Title: Angiomatoid Fibrous Histiocytoma: a Single Institution Case-series
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: AFH
Record Dates: First submitted 2018-11-22; First posted 2018-11-30 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2018-11

CONDITIONS: Angiomatoid Fibrous Histiocytoma
MeSH Terms: conditions — Histiocytoma, Angiomatoid Fibrous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — immunohistochemistry will be performed on FFPE material. EWS-CREB1 and EWS-ATF1 mutation and ALK expression will be analyzed with RT-PCR and/or FISH analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
single institution cases series review of histological and clinical data

DETAILED DESCRIPTION:
single institution cases series review of histological and clinical data Investigators will retrieve from the archives of the Rizzoli Institute all the cases with a histological diagnosis of Angiomatoid Fibrous Histiocytoma. In all cases with enough available material, immunohistochemistry will be performed on slides/formalin-fixed paraffin-embedded tissue tumor material.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients treated at Rizzoli Institute from 01 January 2006 to 31 December 2017
* Diagnosis of Angiomatoid Fibrous Histiocytoma
* Histological slides/formalin-fixed paraffin-embedded tissue tumor (FFPE) blocks from archive available to perform the histology analysis
* Written informed consent prior to any study-specific analysis and/or data collection

Exclusion Criteria:

• Patients with histological diagnosis different from Angiomatoid Fibrous Histiocytoma

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Male and Female with diagnosis of Angiomatoid Fibrous Histiocytoma with histological slides/formalin-fixed paraffin-embedded tissue tumor blocks from archive available to perform the histology analysis
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
selection and review of 9 cases of Angiomatoid Fibrous Histiocytoma | at baseline (Day0)
  investigators will review all the medical records, radiological imaging, and histological slides of all cases to identify the best therapeutic approach.
analysis of EWS-CREB1 and EWS-ATF1 mutation and ALK expression on tissue tumor material | at baseline (Day0)
  In all cases immunohistochemistry will be performed on slides/formalin-fixed paraffin-embedded tissue tumor material. EWS-CREB1 and EWS-ATF1 mutation and ALK expression will be analyzed with RT-PCR and/or FISH analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCC Rizzoli Orthopedic Institute, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
No Individual Patient Data sharing plan has been implemented

REFERENCES:
- [Result] Antonescu CR, Dal Cin P, Nafa K, Teot LA, Surti U, Fletcher CD, Ladanyi M. EWSR1-CREB1 is the predominant gene fusion in angiomatoid fibrous histiocytoma. Genes Chromosomes Cancer. 2007 Dec;46(12):1051-60. doi: 10.1002/gcc.20491. PMID 17724745
- [Result] Bohman SL, Goldblum JR, Rubin BP, Tanas MR, Billings SD. Angiomatoid fibrous histiocytoma: an expansion of the clinical and histological spectrum. Pathology. 2014 Apr;46(3):199-204. doi: 10.1097/PAT.0000000000000073. PMID 24614712
- [Result] Chen G, Folpe AL, Colby TV, Sittampalam K, Patey M, Chen MG, Chan JK. Angiomatoid fibrous histiocytoma: unusual sites and unusual morphology. Mod Pathol. 2011 Dec;24(12):1560-70. doi: 10.1038/modpathol.2011.126. Epub 2011 Aug 5. PMID 21822206
- [Result] Noujaim J, Jones RL, Swansbury J, Gonzalez D, Benson C, Judson I, Fisher C, Thway K. The spectrum of EWSR1-rearranged neoplasms at a tertiary sarcoma centre; assessing 772 tumour specimens and the value of current ancillary molecular diagnostic modalities. Br J Cancer. 2017 Feb 28;116(5):669-678. doi: 10.1038/bjc.2017.4. Epub 2017 Jan 31. PMID 28141799
- [Result] Rossi S, Szuhai K, Ijszenga M, Tanke HJ, Zanatta L, Sciot R, Fletcher CD, Dei Tos AP, Hogendoorn PC. EWSR1-CREB1 and EWSR1-ATF1 fusion genes in angiomatoid fibrous histiocytoma. Clin Cancer Res. 2007 Dec 15;13(24):7322-8. doi: 10.1158/1078-0432.CCR-07-1744. PMID 18094413

DOCUMENTS (1):
  • Study Protocol (2018-09-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT03759327/Prot_000.pdf